CLINICAL TRIAL: NCT02521038
Title: The Use of BRILInta to Optimize ANTiplatelet Therapy (BRILIANT) Registry: The BRILIANT KOREA Registry
Brief Title: Use of Ticagrelor in Korean ACS Patients: The BRILIANT KOREA Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: BK Registry
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — Blood samples for laboratory tests including tests such as, CBC, electrolyte, liver function test, BUN, creatinine, Uric Acid, CRP, Cholesterol panel, etc.
  Urine samples for Urine Analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Brilinta — 90mg bid as a treatment for Acute coronary syndrome. Dose and Duration can be adjusted by the primary physician.

SUMMARY:
Patients with acute coronary syndrome (ACS) require platelet inhibition after treatment. P2Y12 receptor blockage is a well-known, proved method of urgent and effective blockade of the platelet activation, and is applied to the current practice protocol. Ticagrelor is a well-performing P2Y12 receptor blocking agent which is used in these patients. In the same matter, it is essential to prescribe the exact dosage to optimize efficacy within the safety limits. However current studies are based on Western countries, whereas there has been no Ticagrelor patient registry in East-Asia. Thus it is reasonable to study the use of Ticagrelor in a large registry of Korean ACS patients.

The BK registry is a Prospective, Open-label, Multi-center, Real world, Registry, with prospective registration of patients receiving the medication, Ticagrelor. All subjects are to be followed up for 18 months after diagnosis and treatment for ACS.

The purpose of this study is to observe and register clinical data including Major Adverse Cardiovascular Endpoints and any total bleeding occurrence in Korean ACS patients treated with Ticagrelor during 18 month follow-up. Also, the purpose includes to determine compliance of Ticagrelor during post-approval commercial use and to determine prescription pattern of Ticagrelor during post-approval commercial use.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures. Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.
2. Patients who are taking ticagrelor and acetylsalicylic acid daily or Patients who are taking ticagrelor only according to label. All treatment modalities for Acute coronary syndrome (invasive and non-invasive) are allowed.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACS pateints who use Brilinta as a anti-platelet agent
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 'Major Adverse Cardiovascular endpoints' | 18 months
  'Major Adverse Cardiovascular endpoints' assessment will be recorded as number of participants with 'Major Adverse Cardiovascular endpoints'. This measure is a composite outcome, which includes cardiovascular death, myocardial infarction, stroke, stent thrombosis.
Number of participants with Bleeding events | 18 months
  Bleeding event assessment will be recorded as number of participants with Bleeding events. Assessment will be done by the investigator(s) at each routine out-patient follow-up period. Bleeding events will be analyzed according to the 'PLATO bleeding criteria'.

SECONDARY OUTCOMES:
Compliance of Brilinta | 12 months
  Compliance assessment will be recorded as 'taken pills per prescribed pills'. This will be assessed by history taking, self-reports of pill counts. Reports from the 'Korean Health Insurance Review & Assessment Service' can be used to assess the patients' compliance, by the prescription refill rate. Assessment will be done by the investigator(s) at each routine out-patient follow-up period.
Duration of prescribed Brilinta | 12 months
  'Duration of prescribed Brilinta' assessment will be recorded as 'months', which is the actual period Brilinta is prescribed. This will be assessed by hospital records of Brilinta prescriptions. Reports from the 'Korean Health Insurance Review & Assessment Service' can be used to assess the prescription refill rate.
Dosage of prescribed Brilinta | 12 months
  'Dosage of prescribed Brilinta' assessment will be recorded as 'mg', which is the actual dosage Brilinta is prescribed. This will be assessed by hospital records of Brilinta prescriptions. Reports from the 'Korean Health Insurance Review & Assessment Service' can be used to assess the prescription.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Mahaffey KW, Held C, Wojdyla DM, James SK, Katus HA, Husted S, Steg PG, Cannon CP, Becker RC, Storey RF, Khurmi NS, Nicolau JC, Yu CM, Ardissino D, Budaj A, Morais J, Montgomery D, Himmelmann A, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor effects on myocardial infarction and the impact of event adjudication in the PLATO (Platelet Inhibition and Patient Outcomes) trial. J Am Coll Cardiol. 2014 Apr 22;63(15):1493-9. doi: 10.1016/j.jacc.2014.01.038. Epub 2014 Feb 19. PMID 24561148
- [Background] Wallentin L, Lindholm D, Siegbahn A, Wernroth L, Becker RC, Cannon CP, Cornel JH, Himmelmann A, Giannitsis E, Harrington RA, Held C, Husted S, Katus HA, Mahaffey KW, Steg PG, Storey RF, James SK; PLATO study group. Biomarkers in relation to the effects of ticagrelor in comparison with clopidogrel in non-ST-elevation acute coronary syndrome patients managed with or without in-hospital revascularization: a substudy from the Prospective Randomized Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2014 Jan 21;129(3):293-303. doi: 10.1161/CIRCULATIONAHA.113.004420. Epub 2013 Oct 29. PMID 24170388
- [Background] Bansilal S, Bonaca MP, Sabatine MS. Ticagrelor for acute coronary syndromes. Expert Rev Cardiovasc Ther. 2013 Nov;11(11):1473-84. doi: 10.1586/14779072.2013.839205. Epub 2013 Oct 23. PMID 24147518
- [Background] Steg PG, Harrington RA, Emanuelsson H, Katus HA, Mahaffey KW, Meier B, Storey RF, Wojdyla DM, Lewis BS, Maurer G, Wallentin L, James SK; PLATO Study Group. Stent thrombosis with ticagrelor versus clopidogrel in patients with acute coronary syndromes: an analysis from the prospective, randomized PLATO trial. Circulation. 2013 Sep 3;128(10):1055-65. doi: 10.1161/CIRCULATIONAHA.113.002589. Epub 2013 Jul 30. PMID 23900047
- [Background] Berger JS. Aspirin, clopidogrel, and ticagrelor in acute coronary syndromes. Am J Cardiol. 2013 Sep 1;112(5):737-45. doi: 10.1016/j.amjcard.2013.04.055. Epub 2013 Jun 7. PMID 23751937
- [Background] Montalescot G, Lassen JF, Hamm CW, Lapostolle F, Silvain J, ten Berg JM, Cantor WJ, Goodman SG, Licour M, Tsatsaris A, van't Hof AW. Ambulance or in-catheterization laboratory administration of ticagrelor for primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: rationale and design of the randomized, double-blind Administration of Ticagrelor in the cath Lab or in the Ambulance for New ST elevation myocardial Infarction to open the Coronary artery (ATLANTIC) study. Am Heart J. 2013 Apr;165(4):515-22. doi: 10.1016/j.ahj.2012.12.015. Epub 2013 Feb 13. PMID 23537967
- [Background] Wittfeldt A, Emanuelsson H, Brandrup-Wognsen G, van Giezen JJ, Jonasson J, Nylander S, Gan LM. Ticagrelor enhances adenosine-induced coronary vasodilatory responses in humans. J Am Coll Cardiol. 2013 Feb 19;61(7):723-7. doi: 10.1016/j.jacc.2012.11.032. Epub 2013 Jan 9. PMID 23312702